CLINICAL TRIAL: NCT00365508
Title: Comparing the Lozenge to the Patch for Smoking Cessation
Brief Title: Counseling and Nicotine Replacement Therapy in Helping Adult Smokers Quit Smoking
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Fox Chase Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000491296; FCCC-FCRB-04-003-P (Other: Community Clinical Oncology Program Network); 05-818 (Other: Fox Chase Cancer Center)
Record Dates: First submitted 2006-08-16; First posted 2006-08-17 (Estimated); Results first posted 2013-01-30 (Estimated); Last update posted 2016-03-29 (Estimated); Status verified 2016-03

CONDITIONS: Bladder Cancer; Cervical Cancer; Esophageal Cancer; Gastric Cancer; Head and Neck Cancer; Kidney Cancer; Leukemia; Liver Cancer; Lung Cancer; Pancreatic Cancer; Tobacco Use Disorder
Keywords: bladder cancer; cervical cancer; esophageal cancer; gastric cancer; renal cell carcinoma; adult primary liver cancer; non-small cell lung cancer; small cell lung cancer; pancreatic cancer; hypopharyngeal cancer; laryngeal cancer; lip and oral cavity cancer; nasopharyngeal cancer; oropharyngeal cancer; paranasal sinus and nasal cavity cancer; adult acute myeloid leukemia; tongue cancer; tobacco use disorder
MeSH Terms: conditions — Urinary Bladder Neoplasms; Uterine Cervical Neoplasms; Esophageal Neoplasms; Stomach Neoplasms; Head and Neck Neoplasms; Kidney Neoplasms; Leukemia; Liver Neoplasms; Lung Neoplasms; Pancreatic Neoplasms; Tobacco Use Disorder; Carcinoma, Renal Cell; Carcinoma, Hepatocellular; Carcinoma, Non-Small-Cell Lung; Small Cell Lung Carcinoma; Hypopharyngeal Neoplasms; Laryngeal Neoplasms; Mouth Neoplasms; Nasopharyngeal Neoplasms; Oropharyngeal Neoplasms; Leukemia, Myeloid, Acute; Tongue Neoplasms | interventions — Tobacco Use Cessation Devices

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm I (Experimental): Participants apply a transdermal nicotine patch at 3 different time periods during weeks 3-14; a higher-dose patch is applied for weeks 3-8, a medium-dose patch is applied for weeks 9-10, and a lower-dose patch is applied for weeks 11-14.
  Interventions: Drug: nicotine patch
- Arm II (Experimental): Participants receive one oral nicotine lozenge every 1-2 hours in weeks 3-8 (≥ 9 lozenges per day), one lozenge every 2-4 hours in weeks 9-11 (≥ 5 lozenges per day), and 1 lozenge every 4-8 hours in weeks 12-14 (≥ 3 lozenges per day).
  Interventions: Drug: nicotine lozenge

INTERVENTIONS:
Drug: nicotine lozenge — nicotine lozenge
  Arms: Arm II
Drug: nicotine patch — transdermal nicotine patch
  Other Names: transdermal nicotine patch
  Arms: Arm I

SUMMARY:
RATIONALE: Stop-smoking plans, including counseling and nicotine replacement therapy, may help smokers quit smoking. It is not yet known whether counseling and the nicotine lozenge is more effective than counseling and the nicotine patch in helping adult smokers quit smoking.

PURPOSE: This randomized phase III trial is studying counseling and the nicotine lozenge to see how well they work compared to counseling and the nicotine patch in helping smokers quit smoking.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare the efficacy of behavioral counseling and nicotine-replacement therapy with either oral nicotine lozenge (NL) or transdermal nicotine patch (NP), in terms of promoting rates of smoking cessation (e.g., continued abstinence), in adult smokers.
* Examine the degree to which nicotine replacement therapy (NRT) preference, desire to control NRT dosing, irregular smoking schedules, and desire for oral preoccupation moderates the relative efficacy of NL vs NP in promoting smoking cessation.
* Evaluate the impact of the NL on mediators of smoking cessation (i.e., reduced craving, diminished withdrawal symptoms, cue reactivity, and increased perceived control over withdrawal symptoms).

Secondary

* Compare the rate of compliance with NRT across the 2 treatment arms and examine if compliance rate mediates the effects of NRT on quit rates.
* Examine the potential role of genes related to nicotine dependence such as genes related to nicotine metabolism enzymes (e.g., CYP1A1) or genes related to dopamine concentrations (e.g., DRD2).

OUTLINE: This is a randomized, open-label, multicenter study. Participants are stratified according to study center. Participants are randomized to 1 of 2 intervention arms.

All participants undergo smoking cessation counseling in weeks 1, 3, 5, 7, and 9. Beginning in week 3, participants are asked to quit smoking for 12 weeks (weeks 3-14).

* Arm I: Participants apply a transdermal nicotine patch at 3 different time periods during weeks 3-14; a higher-dose patch is applied for weeks 3-8, a medium-dose patch is applied for weeks 9-10, and a lower-dose patch is applied for weeks 11-14.
* Arm II: Participants receive one oral nicotine lozenge every 1-2 hours in weeks 3-8 (≥ 9 lozenges per day), one lozenge every 2-4 hours in weeks 9-11 (≥ 5 lozenges per day), and 1 lozenge every 4-8 hours in weeks 12-14 (≥ 3 lozenges per day).

The moderating variables (e.g., nicotine replacement-therapy [NRT] preference and the smoker's desire to control NRT dosing) are assessed at baseline. The mediating variables (i.e., reduced craving, diminished withdrawal symptoms, cue reactivity, and increased perceived control over withdrawal symptoms) are assessed at baseline and then at weeks 5, 7, 9, within weeks 14-16, and within weeks 26-28. Continuous abstinence will be measured at week 27.

PROJECTED ACCRUAL: A total of 700 participants will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Smokes at least 10 cigarettes a day on average for the past year
* No prior diagnosis of cancer (unless completed treatment AND no evidence of disease within the past 5 years)
* Able to use nicotine replacement therapy

PATIENT CHARACTERISTICS:

* Able to communicate in English
* Must reside in the geographic area for ≥ 6 months
* Current asthma, ulcer, or diabetes allowed provided medical clearance from the participant's physician is obtained
* No evidence of drug or alcohol abuse
* No known HIV positivity
* No heart disease, including any of the following:

  * Current diagnosis of coronary artery disease
  * Abnormal heart rhythm or an arrhythmia
  * Heart failure
  * Heart valve disease
  * Congenital heart disease
  * Heart muscle disease or cardiomyopathy
  * Pericardial disease
  * Aorta disease
  * Vascular disease
  * Myocardial infarction
  * High blood pressure (defined as blood pressure > 140/90 mm Hg) not receiving antihypertensive medication

    * History of or current high blood pressure controlled by antihypertensive medication and having medical clearance from physician allowed
* No allergy to adhesive tape or latex
* Not pregnant or nursing
* Negative pregnancy test
* Fertile participants must use effective contraception during and for ≥ 1 month prior to and after completion of study treatment

PRIOR CONCURRENT THERAPY:

* At least 30 days since prior and no concurrent benzodiazepine (e.g., diazepam, alprazolam, or lorazepam)
* At least 6 months since prior antiretroviral medications
* At least 6 months since prior and no concurrent medication for depression (e.g., phenelzine sulfate, pargyline hydrochloride, tranylcypromine sulfate, paroxetine hydrochloride, sertraline hydrochloride, fluoxetine hydrochloride)
* No concurrent antipsychotics (e.g., lithium) or theophylline
* No concurrent substance abuse treatment
* No concurrent bupropion hydrochloride
* No other concurrent pharmacologic aid or any other form of formal assistance for smoking cessation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 642 (Actual)
Dates: Start 2006-02; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert A. Schnoll, PhD, Study Chair — Fox Chase Cancer Center - Cheltenham
Locations (10):
- United States (10):
  - Howard University Cancer Center, Washington D.C., District of Columbia
  - CCOP - Mount Sinai Medical Center, Miami Beach, Florida
  - Medical College of Georgia Cancer Center, Augusta, Georgia
  - Fox Chase Virtua Health Cancer Program at Virtua Memorial Hospital Burlington County, Mount Holly, New Jersey
  - Hematology Oncology Associates of Central New York, PC - Northeast Center, East Syracuse, New York
  - Don Monti Comprehensive Cancer Center at North Shore University Hospital, Manhasset, New York
  - Geisinger Cancer Institute at Geisinger Health, Danville, Pennsylvania
  - Fox Chase Cancer Center - Philadelphia, Philadelphia, Pennsylvania
  - CCOP - Main Line Health, Wynnewood, Pennsylvania
  - Nashville General Hospital at Meharry, Nashville, Tennessee

REFERENCES:
- [Derived] Theodoulou A, Fanshawe TR, Leavens E, Theodoulou E, Wu AD, Heath L, Stewart C, Nollen N, Ahluwalia JS, Butler AR, Hajizadeh A, Thomas J, Lindson N, Hartmann-Boyce J. Differences in the effectiveness of individual-level smoking cessation interventions by socioeconomic status. Cochrane Database Syst Rev. 2025 Jan 27;1(1):CD015120. doi: 10.1002/14651858.CD015120.pub2. PMID 39868569

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited through ads/physician referral at: FCCC, Geisinger Medical Center, Hematology Oncology Associates of Central NY, Howard University, LSU, Main Line Health System, Medical College of GA, Meharry Medical College, Mount Sinai Medical Center (Miami), North Shore University, SUNY Downstate Medical Center, and Virtua Health.
Pre-assignment Details: 1299 individuals were screened for this trial over 4 years; 454 individuals were ineligible, 194 refused enrollment, and 651 were randomized. Nine individuals either withdrew from the study prior to treatment or were found to be ineligible after randomization and were removed from the intent-to-treat sample. The final ITT sample was 642 (321/arm).
Groups:
- Nicotine Patch: Participants apply a transdermal nicotine patch at 3 different time periods during weeks 3-14; a higher-dose patch is applied for weeks 3-8, a medium-dose patch is applied for weeks 9-10, and a lower-dose patch is applied for weeks 11-14.
- Nicotine Lozenge: Participants receive one oral nicotine lozenge every 1-2 hours in weeks 3-8 (≥ 9 lozenges per day), one lozenge every 2-4 hours in weeks 9-11 (≥ 5 lozenges per day), and 1 lozenge every 4-8 hours in weeks 12-14 (≥ 3 lozenges per day).
Period: Overall Study
Arm/Group | Nicotine Patch | Nicotine Lozenge
Started | 321 | 321
Completed | 182 | 167
Not Completed | 139 | 154
Not completed — Lost to Follow-up | 139 | 154

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I | Arm II | Total
Number analyzed (Participants) | 321 | 321 | 642
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.7 (12.7) | 44.8 (11.9) | 44.7 (12.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 195 | 170 | 365
  Male | 126 | 151 | 277

OUTCOME MEASURES:

1. Primary Outcome: 24-hour Point Prevalence Abstinence at the 6-month Follow up
Time Frame: 6-months
Population: Intent to treat analysis (lost to follow-up = smoker)
Measure: Number; unit: participants
Arm/Group | Arm I | Arm II
Number analyzed (Participants) | 321 | 321
participants | 50 | 35
Statistical Analysis 1: Comparison: Arm I vs Arm II; Chi-square was used to examine the relationship between treatment arm and 24-hour point prevalence abstinence at 6-months; Test type: Superiority or Other; p = .05, Chi-squared — a priori threshold for statistical significance

2. Secondary Outcome: Rate of Compliance During the First 2 Weeks
Description: Applied to use of the intervention (number of lozenges/day or number of patches used per week) not considering abstinence
Time Frame: 2 weeks
Population: Intent to treat
Measure: Number; unit: participants
Arm/Group | Arm I | Arm II
Number analyzed (Participants) | 321 | 321
participants | 231 | 87

ADVERSE EVENTS:
Time Frame: 6 months
Description: Administered a checklist of side effects from NRT and collected any additional information on adverse events.
Arm/Group | Arm I | Arm II
Serious Adverse Events (participants affected / at risk) | 4/321 | 7/321
Other Adverse Events (participants affected / at risk) | 0/321 | 0/321
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (N=321) | Arm II (N=321)
Stroke (Cardiac disorders) | 2 (2) | 0 (0)
Seizure (Nervous system disorders) | 1 (1) | 1 (1)
killed in car accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Heart disease (Cardiac disorders) | 0 (0) | 1 (1)
ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
appendicitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
heart attack (Cardiac disorders) | 0 (0) | 1 (1)
cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Abcessed tooth (Surgical and medical procedures) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
The study was an effectiveness trial so external vs. internal validity was emphasized. Many participants were lost to follow-up.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No